CLINICAL TRIAL: NCT03291210
Title: Effect of O2 Tension on Myocardial Injury During TAVI
Brief Title: O2 Tension During TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Prinicipal investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAVI-O2
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Troponin
Keywords: hyperoxemia; myocardial injury; transcatheter aortic valve replacement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normoxemia (Experimental): Patients randomized to the normoxemia group receives inspired oxygen fraction of 0.3 from initiation of induction of anesthesia to the end of the procedure.
  Interventions: Other: normal inspired oxygen fraction
- Hyperoxemia (Active Comparator): Patients randomized to the hyperoxemia group receives inspired oxygen fraction of 0.8 from initiation of induction of anesthesia to the end of the procedure.
  Interventions: Other: high inspired oxygen fraction

INTERVENTIONS:
Other: normal inspired oxygen fraction — receives inspired oxygen fraction of 0.3
  Arms: Normoxemia
Other: high inspired oxygen fraction — receives inspired oxygen fraction of 0.8
  Arms: Hyperoxemia

SUMMARY:
Hyperoxemia can produce various complications including oxidative stress and myocardial injury. We hypothesized that the normoxic group would have lower myocardial injury compared to hyperoxic group after transcatheter aortic valve replacement.

DETAILED DESCRIPTION:
Hyperoxemia can produce various complications, such as excessive oxidative stress, hyperoxia-induced vasoconstriction, increased perfusion heterogeneity, and resultant myocardial injury. Previous studies have been observed higher mortality in patient group maintained with supranormal oxygenation after resuscitation from cardiac arrest. However, the effect of hyperoxia vs. normoxia on myocardial injury during transcatheter aortic valve replacement (TAVR) has not been well investigated. We hypothesized that the normoxic group would have lower myocardial injury compared to hyperoxic group after TAVR.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for transcatheter aortic valve replacement due to aortic stenosis

Exclusion Criteria:

* Transapical approach
* Pre-procedural PaO2 < 65 mmHg or oxygen support therapy
* Pre-procedural severe kidney injury (end-stage renal disease)
* Pre-procedural chronic pulmonary disease, symptomatic asthma
* Pre-procedural Tb-destroyed lung
* Lung cancer
* History of acute coronary syndrome within 6 months
* Pre-procedural elevated Troponin I or CKMB
* History of stroke or transient ischemic attack within 6 months
* Refuse to participate
* Pregnant

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Troponin I | 72 hours after the end of procedure
  Area under the curve of troponin I

SECONDARY OUTCOMES:
CK MB | 72 hours after the end of procedure
  Area under the curve of CK MB
Changes in cerebral oximetry | through procedure completion, an average of 3 hours
  changes in cerebral oximetry during the procedure
Delirum | through admission completion, an average of 5 days
  Newly onset delirium
AKI or RRT | through admission completion, an average of 5 days
  Newly onset acute kidney injury or renal replacement therapy
stroke, myocardial infarction or mortality | through admission completion, an average of 5 days
  Newly onset stroke, myocardial infarction or mortality

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided